CLINICAL TRIAL: NCT04191486
Title: A Phase 2 Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of T-817MA in Patients With Mild Cognitive Impairment Due to Alzheimer's Disease or Mild Alzheimer's Disease
Brief Title: Efficacy and Safety of T-817MA in Patients With Mild Cognitive Impairment Due to Alzheimer's Disease (AD) or Mild AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: FUJIFILM Toyama Chemical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T817MAEU201; 2018-003567-66 (EudraCT Number)
Record Dates: First submitted 2019-11-26; First posted 2019-12-09 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-02

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — 1-(3-(2-(1-benzothiophen-5-yl) ethoxy) propyl)-3-azetidinol maleate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T-817MA (448 mg) (Experimental)
  Interventions: Drug: T-817MA
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: T-817MA — 224mg T-817MA orally once daily for first 4 weeks, and then 448mg T-817MA orally once daily for the following weeks.
  Arms: T-817MA (448 mg)
Drug: Placebo — Placebo once daily
  Arms: Placebo

SUMMARY:
Primary objective is to evaluate the neuroprotective effect of T-817MA on Tau protein phosphorylated at threonine 181 (p-tau 181) in cerebrospinal fluid (CSF) compared with placebo in patients with a diagnosis of MCI due to AD or mild AD.

Secondary objectives are:

1. To evaluate in patients on T-817MA and placebo:

   * cognitive function measured by the Clinical Dementia Rating Scale Sum of Boxes (CDR-sb) and working memory and attention domain as measured by the Cognitive Functional Composite (CFC).
   * AD-related biomarkers in CSF and plasma
   * imaging analysis using volumetric magnetic resonance imaging (vMRI)
   * alpha/theta ratio of the electroencephalogram (EEG)
2. To evaluate the safety of T-817MA by clinical laboratory tests and adverse events (AEs).
3. To evaluate the pharmacokinetics of T-817MA

ELIGIBILITY:
Key Inclusion Criteria:

* Female of non-childbearing potential or male, ages 50 to 80 years (inclusive)
* MCI due to AD or mild AD per NIA-AA diagnostic criteria (Jack et al., 2018), with MMSE 24 to 30 (inclusive)
* CSF results at Screening consistent with the presence of Aß and p-tau181 abnormality (≤1000 pg/ml for Aß, ≥19 pg/ml for p-tau181).
* Taking stable dose of AChE Inhibitor (donepezil, galantamine or rivastigmine) at least for 3 months prior to randomization, or not taking any AChE Inhibitors.

Key Exclusion Criteria:

* MRI of the brain within the previous 2 years that showed pathology that would be inconsistent with a diagnosis of AD
* Taking memantine
* Any contraindications to lumbar puncture
* Any contraindications to MRI

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — If male, patients must:
  1. agree he will not donate sperm during the study and until 104 days after the last dose, AND
  2. be required to use highly effective methods of contraception during the study and until 104 days after the last dose
  If female, patients must:
  1. be post-menopausal (i.e. no menses for 12 months without an alternative medical cause) OR
  2. be permanently sterilized with methods including hysterectomy, bilateral salpingectomy and bilateral oophorectomy
Enrollment: 221 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
The change in the CSF p-tau181 from Baseline to Week 78 | Baseline to Week 78

SECONDARY OUTCOMES:
The change in the CSF p-tau181 from Baseline to Week 52 | Baseline to Week 52
The change in the CSF p-tau217 from Baseline to Weeks 52 and 78 | Baseline to Weeks 52 and 78
The change in the CSF total tau from Baseline to Weeks 52 and 78 | Baseline to Weeks 52 and 78
The change in the CSF Aβ1-42 from Baseline to Weeks 52 and 78 | Baseline to Weeks 52 and 78
The change in the CSF Aβ1-40 from Baseline to Weeks 52 and 78 | Baseline to Weeks 52 and 78
The change in the CSF neurofilament light (NFL) from Baseline to Weeks 52 and 78 | Baseline to Weeks 52 and 78
The change in the CSF neurogranin from Baseline to Weeks 52 and 78 | Baseline to Weeks 52 and 78
The change in the CSF YKL-40 from Baseline to Weeks 52 and 78 | Baseline to Weeks 52 and 78
The change in the CSF Aβ1-42/Aβ1-40 ratio from Baseline to Weeks 52 and 78 | Baseline to Weeks 52 and 78
The change in the plasma Aβ1-42 from Baseline to Weeks 52 and 78 | Baseline to Weeks 52 and 78
The change in the plasma Aβ1-40 from Baseline to Weeks 52 and 78 | Baseline to Weeks 52 and 78
The change in the plasma NFL from Baseline to Weeks 52 and 78 | Baseline to Weeks 52 and 78
The change in cognitive function assessed by CDR-sb and working memory and attention domain as measured by the CFC from Baseline to Weeks 28, 52 and 78 | Baseline to Weeks 28, 52 and 78
The change in brain volume (total brain volume (TBV), ventricular volume and hippocampal volume) and cortical thickness measured by vMRI from Baseline to Weeks 52 and 78 | Baseline to Weeks 52 and 78
The change in alpha/theta ratio measured by the EEG from Baseline to Weeks 52 and 78 | Baseline to Weeks 52 and 78
Safety as assessed by the occurrence of AEs, clinical laboratory tests, vital signs, physical examinations, ECGs | Screening to Week 82
Population PK analysis of T-817MA with assessment of maximum plasma concentration (Cmax) | Weeks 16, 28, 40, and 65
Population PK analysis of T-817MA with assessment of minimum plasma concentration (Cmin) | Weeks 16, 28, 40, and 65
Population PK analysis of T-817MA with assessment of total daily exposure (AUC0-24h) | Weeks 16, 28, 40, and 65

CONTACTS AND LOCATIONS:
Overall Officials: Philip Scheltens, MD, PhD, Study Director — VUmc Alzheimer Centrum
Locations (37):
- Czechia (5):
  - FNUSA - Mezinarodni centrum klinickeho vyzkumu, Brno
  - FNHK - Neurologicka klinika, Hradec Králové
  - A-shine, s.r.o., Pilsen
  - CLINTRIAL, s.r.o., Prague
  - VESTRACLINICS, s.r.o., Rychnov
- Germany (9):
  - Klinik für Psychiatrie, Psychosomatik und Psychotherapie Universitätsklinikum Frankfurt, Frankfurt
  - Klinik für Neurologie Universitätsklinikum Schleswig-Holstein, Kiel
  - Klinik und Poliklinik für Neurologie Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Magdeburg Institut für Kognitive Neurologie und Demenzforschung, Magdeburg
  - Institut für Studien zur Psychischen Gesundheit (ISPG), Mannheim
  - Technische Universität München, München
  - Universitätsklinikum Münster Klinik für Allgemeine Neurologie, Münster
  - Universitätsmedizin Rostock Zentrum für Nervenheilkunde Klinik für Psychosomatik und Psychotherapeutische Medizin, Rostock
  - Universitätsklinikum Ulm Studienzentrum Klinik für Neurologie, Ulm
- Hungary (4):
  - Debreceni Egyetem KK, Pszichiátriai Klinika, Budapest
  - Jávorszky Ödön Városi Kórház, Gyógyszertár, Debrecen
  - Semmelweis Egyetem, Pszichiátriai és Pszichoterápiás Klinika, Győr
  - Semmelweis Egyetem Neurológiai Klinika Gyógyszertára, C földszint, Vác
- Ireland (2):
  - St. Vincent's University Hospital, Dublin
  - Tallaght University Hospital., Dublin
- Netherlands (4):
  - Brain Research Center Den Bosch, 's-Hertogenbosch
  - Brain Research Center, Amsterdam
  - Amphia ziekenhuis, Breda
  - Isala ziekenhuis, Zwolle
- Spain (8):
  - Hospital General Universitari d' Elx, Alicante
  - Fundació ACE, Barcelona
  - Àrea Gestió Documentació Assaigs Clínics-AGDAC Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Clínico Universitario Virgen de La Arrixaca, El Palmar
  - CAE Oroitu, Getxo
  - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Victoria Eugenia - Cruz Roja, Seville
  - Hospital Viamed Montecanal, Zaragoza
- United Kingdom (5):
  - University of Bath, Bath
  - Southmead Hospital North Bristol NHS Trust, Bristol
  - Glasgow memory Clinic, Glasgow
  - Imperial College Healthcare NHS Trust, London
  - Memory Assessment & Research Centre, Southampton

IPD SHARING:
Plan to Share IPD: Undecided
Details for sharing data have not been decided yet.